CLINICAL TRIAL: NCT01342900
Title: Intraoperative Monitoring and Optimisation of Tissue Oxygenation In High-Risk Surgical Patients for Reduction of Postoperative Complications: a Pilot Study
Brief Title: Intraoperative Optimisation of Tissue Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof.dr.T.W.L.Scheeren, Prof.dr., University Medical Center Groningen
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: IOTO-001
Record Dates: First submitted 2011-04-21; First posted 2011-04-27 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Higk Risk Surgery
Keywords: tissue oxygenation; higk risk surgery; high risk patient; postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard care (No Intervention): The data from the InSPectra Monitor in the Control group will be inaccessible for the Investigator since this is not a part of their daily medical practice
- Treatment group, (Active Comparator): The data given by the monitor will be available for the Investigator and used to apply the optimization protocol
  Interventions: Device: connected to the InSpectra Monitor

INTERVENTIONS:
Device: connected to the InSpectra Monitor
  Arms: Treatment group,

SUMMARY:
Monitoring and optimizing tissue oxygenation (StO2) in high-risk surgery and/or high-risk surgical patients may decrease the risk of postoperative complications.

Tissue hypoxia occurs frequently during high-risk surgery in high-risk patients. The investigators want to see if an algorithm aimed at optimizing intraoperative tissue oxygenation reduces perioperative complications as well as length of stay in the intensive care unit (ICU LOS), 28-day mortality, and the duration of mechanical ventilation in these patients.

ELIGIBILITY:
Inclusion Criteria:

. Major elective surgery

* Aged over 65 years with moderate functional limitation of one or more organ systems
* ASA classification III or IV, i.e. severe cardiac, vascular, respiratory or metabolic illness resulting in severe functional limitation
* Routine use of arterial and central venous lines
* Planned postoperative stay on ICU or PACU

Exclusion Criteria:

* Refusal of consent
* acute myocardial ischemia prior to enrolment
* patients receiving palliative treatment only
* disseminated malignancy
* patients unlikely to survive more than 6 hours
* emergency surgery
* transplantations
* neurosurgical patients
* patients undergoing extensive liver surgery requiring low CVP management

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
incidence of perioperative complications | during operation
  organ dysfunction, SOFA score, troponin T, creatinin, CRP

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W.L. Scheeren, Prof.dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] van Beest PA, Vos JJ, Poterman M, Kalmar AF, Scheeren TW. Tissue oxygenation as a target for goal-directed therapy in high-risk surgery: a pilot study. BMC Anesthesiol. 2014 Dec 16;14:122. doi: 10.1186/1471-2253-14-122. eCollection 2014. PMID 25580087